CLINICAL TRIAL: NCT05130528
Title: Therapeutic Intervention Supporting Development From the Neonatal Intensive Care Unit to 6 Months for Infants Post Hypoxic-Ischemic Encephalopathy
Brief Title: Therapeutic Intervention Supporting Development From NICU to 6 Months for Infants Post Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Barbara Sargent, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHLA-21-00290; P2CHD101912 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2021-11-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Hypoxic-Ischemic Encephalopathy
Keywords: infant
MeSH Terms: conditions — Cerebral Palsy; Hypoxia-Ischemia, Brain | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Infants randomly assigned to this arm will not receive any study intervention but will continue with any intervention in the community recommended by their health care team.
- Sensorimotor Intervention (Experimental): Infants randomly assigned to this arm will participate in the sensorimotor intervention starting in the hospital and lasting for 6 months. This intervention includes 10 visits with a physical or occupational therapist and parent working together to advance an intervention program and 6 months of parent daily intervention. In addition, this arm will continue with any intervention in the community recommended by their health care team.
  Interventions: Behavioral: Sensorimotor Intervention

INTERVENTIONS:
Behavioral: Sensorimotor Intervention — Infants in the experimental group will receive 2 sensorimotor intervention sessions in the Neonatal Intensive Care Unit (NICU) and 8 sensorimotor intervention sessions in the home or in a clinic (parent choice) at 1, 3, 5, 8, 11, 15, 20, 26 weeks post NICU discharge. The 2 intervention sessions in the NICU will consist of collaborating with parents to recognize their infant's cues to engage in interaction, readiness for sensory exposures, and anticipatory guidance on the transition to home. The 8 intervention sessions in the home will focus on supporting the parents to read their infant's cues to identify the ideal times for interaction and provide 20 minutes of daily intervention addressing four key principles: encourage 1) self-initiated movement, 2) movement variability, 3) visual and manual object interaction, and 4) social interaction. Parents are encouraged not to impose movement on the infant but to encourage movement through environmental enrichment
  Other Names: Supporting and Enhancing NICU Sensory Experiences (SENSE); Supporting Play, Exploration, and Early Developmental Intervention (SPEEDI)
  Arms: Sensorimotor Intervention

SUMMARY:
The purpose of this study is to evaluate the feasibility and begin to evaluate the effect of a sensorimotor intervention (SMI) provided in the first 6 months of life for infants with hypoxic-ischemic encephalopathy.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a form of newborn brain injury resulting from a lack of oxygen or blood flow to the brain. Over 85 percent of infants with HIE now survive to discharge from the Neonatal Intensive Care Unit (NICU). Therapeutic hypothermia, now standard of care for HIE, improves survival, but does not decrease the incidence of moderate-severe disability or cerebral palsy. Therefore, infants with HIE may benefit from close developmental surveillance and a sensorimotor intervention that may induce positive neuroplasticity and optimize developmental outcomes. In addition, parents of infants with HIE may benefit from anticipatory guidance to promote global development and extensive education on how to monitor their infant for neurological signs and developmental delays that would warrant further medical and therapeutic assessments and services.

The purpose of this study is to evaluate the feasibility and begin to evaluate the effect of a sensorimotor intervention (SMI) provided in the first 6 months of life. Twenty infants with moderate or severe HIE will be recruited and randomized into one of two groups: 1) standard care, and 2) standard care plus SMI. Infants in the SMI group will receive 2 intervention sessions in the NICU and 8 sessions in the home from 1 week to 6 months post discharge. The SMI will focus on supporting parents' ability to enhance motor-based problem solving and global development during the transition from NICU to home. Through this combined parent and therapist support intervention, the parents are empowered to provide their infants daily opportunities for sensorimotor play, increasing the likelihood of developmental change.

Outcomes will be measured at baseline, NICU discharge, and at 3 months and 6 months of age. Feasibility of enrolling, implementing the interventions, and completing the measurement model will be assessed. Secondary outcomes will include standardized assessments of motor and cognitive development of the infants and standardized assessments of confidence and stress of the parents. In addition, baseline neuroimaging data and the results of tests to detect cerebral palsy at 3 and 6 months of age will be used to characterize the participants and will be analyzed as potential moderators of treatment effects in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Infants with moderate or severe hypoxic-ischemic encephalopathy (HIE) based on the modified Sarnat Exam on admission and has started to receive therapeutic hypothermia for 72 hours.
* Cared for in the Newborn and Infant Critical Care Unit (NICCU) at Children's Hospital Los Angeles (CHLA).
* Family lives within 60 miles of CHLA.
* One parent/legal guardian has provided signed and dated informed consent form agreeing to the child's participation and the parent's own participation.

Exclusion Criteria:

* Infant born preterm.
* Infant with congenital anomalies, chromosomal or microarray abnormalities.
* Infant with microcephaly.
* Infants who have been redirected for comfort care.
* Infants who are medically unstable.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Neonatal Intensive Care Unit component of the intervention. | 2 weeks
  Feasibility will be defined as the proportion of parent/infant dyads completing 2 assessments and 2 parent/therapist collaborative sensorimotor intervention sessions before Neonatal Intensive Care Unit discharge.
Feasibility of the entire sensorimotor intervention. | 6 months
  Feasibility will be defined as: (a) the proportion of parent/infant dyads completing 80% or more of the recommended 10 sensorimotor intervention sessions, and (b) the parents reporting daily completion of the sensorimotor intervention on 80% of randomly sampled days.

SECONDARY OUTCOMES:
Test of Infant Motor Performance (TIMP) | 3 months
  Standardized motor assessment for infants less than 4 months of age; raw scores will be used to document change over time.
Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4): fine motor, gross motor and cognitive scaled scores | 6 months
  Standardized developmental assessment; scaled scores for the fine motor, gross motor, and cognitive subtests will be used to document change over time.
Sensory Profile 2 (SP2) | 3 months, 6 months
  Standardized questionnaire that assesses the infant's sensory system.
Maternal Confidence Questionnaire (MCQ) | 3 months, 6 months
  Standardized questionnaire that assesses maternal confidence in parenting.
Parent Stress Index - Short Form (PSI-sf) | 3 months, 6 months
  Standardized questionnaire that assesses the level of stress associated with the parenting role.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C Dusing, PhD, PT, Principal Investigator — University of Southern California / Children's Hospital Los Angeles; Barbara Sargent, PhD, PT, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No